CLINICAL TRIAL: NCT01379209
Title: A Phase 1/2a, Open-Label, Multicenter, Dose-Escalation Study to Evaluate the Safety and Tolerability of Intravenous Administration of RGI-2001 in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation (AHSCT)
Brief Title: Intravenous Administration of RGI-2001 in Patient Undergoing Allogenic Hematopoietic Stem Cell Transplantation (AHSCT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RGI-2001-02
Record Dates: First submitted 2011-06-17; First posted 2011-06-23 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-09

CONDITIONS: Graft Versus Host Disease
Keywords: AHSCT; Bone Marrow Transplant; Leukemia; myelodysplastic syndrome; hematological malignancies; Graft-versus-host-disease; GvHD; Hematopoietic Stem Cell Transplantation; Stem Cell; Transplantation
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Hematologic Neoplasms | interventions — KRN 7000; Calcineurin Inhibitors; Transplantation Conditioning; Methotrexate; Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- RGI-2001 0.001 μg/kg + Standard of Care GVHD Prophylaxis (Experimental): RGI-2001 will be add to standard treatment with a calcineurin inhibitor, in combination with either methotrexate, mycophenolate mofetil, or sirolimus all at doses as per the institutional protocols
  Dose escalation cohort 1 in part 1 of this study will include 2-6 patients
  Interventions: Drug: RGI-2001; Drug: Calcineurin Inhibitors; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Conditioning Regimen; Procedure: Allogeneic Bone Marrow Transplantation; Drug: Methotrexate; Drug: Mofetil Mycophenolate; Drug: sirolimus
- RGI-2001 0.01 μg/kg + Standard of Care GVHD Prophylaxis (Experimental): RGI-2001 will be add to standard treatment with a calcineurin inhibitor, in combination with either methotrexate, mycophenolate mofetil, or sirolimus all at doses as per the institutional protocols
  Cohort 2 in part 1 of this study will include 2-6 patients
  Interventions: Drug: RGI-2001; Drug: Calcineurin Inhibitors; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Conditioning Regimen; Procedure: Allogeneic Bone Marrow Transplantation; Drug: Methotrexate; Drug: Mofetil Mycophenolate; Drug: sirolimus
- RGI-2001 0.1 μg/kg + Standard of Care GVHD Prophylaxis (Experimental): RGI-2001 will be add to standard treatment with a calcineurin inhibitor, in combination with either methotrexate, mycophenolate mofetil, or sirolimus all at doses as per the institutional protocols
  Cohort 3 in part 1 of this study will include 2-6 patients
  Interventions: Drug: RGI-2001; Drug: Calcineurin Inhibitors; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Conditioning Regimen; Procedure: Allogeneic Bone Marrow Transplantation; Drug: Methotrexate; Drug: Mofetil Mycophenolate; Drug: sirolimus
- RGI-2001 1.0 μg/kg + Standard of Care GVHD Prophylaxis (Experimental): RGI-2001 will be add to standard treatment with a calcineurin inhibitor, in combination with either methotrexate, mycophenolate mofetil, or sirolimus all at doses as per the institutional protocols
  Cohort 4 in part 1 of this study will include 2-6 patients
  Interventions: Drug: RGI-2001; Drug: Calcineurin Inhibitors; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Conditioning Regimen; Procedure: Allogeneic Bone Marrow Transplantation; Drug: Methotrexate; Drug: Mofetil Mycophenolate; Drug: sirolimus
- RGI-2001 10 μg/kg + Standard of Care GVHD Prophylaxis (Experimental): RGI-2001 will be add to standard treatment with a calcineurin inhibitor, in combination with either methotrexate, mycophenolate mofetil, or sirolimus all at doses as per the institutional protocols
  Cohort 5 in part 1 of this study will include 2-6 patients
  Interventions: Drug: RGI-2001; Drug: Calcineurin Inhibitors; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Conditioning Regimen; Procedure: Allogeneic Bone Marrow Transplantation; Drug: Methotrexate; Drug: Mofetil Mycophenolate; Drug: sirolimus
- RGI-2001 100 μg/kg + Standard of Care GVHD Prophylaxis (Experimental): RGI-2001 will be add to standard treatment with a calcineurin inhibitor, in combination with either methotrexate, mycophenolate mofetil, or sirolimus all at doses as per the institutional protocols
  Cohort 6 in part 1 of this study will include 2-6 patients
  Interventions: Drug: RGI-2001; Drug: Calcineurin Inhibitors; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Conditioning Regimen; Procedure: Allogeneic Bone Marrow Transplantation; Drug: Methotrexate; Drug: Mofetil Mycophenolate; Drug: sirolimus
- RGI-2001 250μg/kg + Standard of Care GVHD Prophylaxis (Experimental): RGI-2001 will be add to standard treatment with a calcineurin inhibitor, in combination with either methotrexate, mycophenolate mofetil, or sirolimus all at doses as per the institutional protocols
  Cohort 7 in part 1 of this study will include 2-6 patients (optional)
  Interventions: Drug: RGI-2001; Drug: Calcineurin Inhibitors; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Conditioning Regimen; Procedure: Allogeneic Bone Marrow Transplantation; Drug: Methotrexate; Drug: Mofetil Mycophenolate; Drug: sirolimus
- RGI-2001 + Standard of Care GVHD Prophylaxis (Experimental): RGI-2001 will be add to standard treatment with a calcineurin inhibitor, in combination with either methotrexate, mycophenolate mofetil, or sirolimus all at doses as per the institutional protocols
  In part 2 of this study the best dose or doses determined from part 1 will be administered in up to 30 persons.
  Interventions: Drug: RGI-2001; Drug: Calcineurin Inhibitors; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Conditioning Regimen; Procedure: Allogeneic Bone Marrow Transplantation; Drug: Methotrexate; Drug: Mofetil Mycophenolate; Drug: sirolimus

INTERVENTIONS:
Drug: RGI-2001 — A single administration of RGI-2001 on Day 0 post AHSCT.
  Other Names: KRN-7000; RGI-7000
Drug: Calcineurin Inhibitors — GVHD prophylaxis according to institutional guidelines. Subjects could have received any number/combinations of treatments.
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — According to institutional guidelines.
Drug: Conditioning Regimen — Myeloablative preparative treatment according to institutional guidelines. Subjects could have received any number/combinations of treatments.
Procedure: Allogeneic Bone Marrow Transplantation — According to institutional guidelines
Drug: Methotrexate
  Other Names: Administered for GVHD prophylaxis as per institutional guidelines
Drug: Mofetil Mycophenolate
  Other Names: Administered for GVHD prophylaxis as per institution guidelines
Drug: sirolimus — Administered for GVHD prophylaxis as per institutional guidelines

SUMMARY:
The clinical trial is a Phase 1/2a, open-label, multi-center, dose-escalation study to evaluate the safety, tolerability and pharmacokinetic profile of RGI-2001 in patients undergoing AHSCT, with radiation or non-radiation myeloablative preparative treatment.

The study will be separated into two parts; a dose escalation phase to assess safety, followed by a large expansion phase to further evaluate the pharmacologic effects of either a Maximum Tolerated Dose, Maximum Feasible Dose or optimal pharmacologically active dose of RGI-2001. The initial dose escalation safety portion of the study (Part 1) will include higher risk patients and limit the unrelated donor transplants. After safety is established in part 1 of the study, the second portion of the study will expand the enrollment criteria and allow transplantation by either related or unrelated donors.

This study will endeavor to identify the dose range at which RGI-2001 has an acceptable safety profile, at which biologic activity is observed, and to guide possible dose levels to utilize in later phase studies based on biological activity.

DETAILED DESCRIPTION:
The clinical trial is a Phase 1/2a, open-label, multi-center, dose-escalation study to evaluate the safety, tolerability and pharmacokinetic profile of RGI-2001 in patients undergoing AHSCT, with radiation or non-radiation myeloablative preparative treatment.

In Part 1 (Phase 1: Dose Escalation Phase), patients will receive a single intravenous administration of RGI-2001 approximately 30 minutes after completion of the transplant (either allogeneic PBSCs or allogenic bone marrow transplantation (unmodified)) with the dosage based upon the assigned treatment cohort. Eligible patients will be enrolled in five to seven centers in the United States. Patients who are undergoing AHSCT will be enrolled in a sequential group dose-escalating fashion to determine the safety, tolerability, pharmacokinetic profile, and the MTD or MFD of RGI-2001. It is anticipated that up to six dose levels will be evaluated in Part 1, with an option for an additional cohort (Cohort 7) if the MTD is not reached and pharmacodynamic markers suggest higher doses are warranted.

In Part 2 (Expansion Phase), one or more doses below the MTD or MFD will be selected based on a potential correlation between GvHD and biological activity to further assess safety and biologic activity. Approximately 30 patients who are undergoing either allogeneic PBSCs or allogenic bone marrow transplantation (unmodified) will be enrolled in Part 2 of the study.

Patients will be monitored for safety for 29 days after the transplant procedure.

All patients will be followed for 100 days following transplant procedure for the incidence of acute GvHD, according to the Modified Keystone Criteria for grading acute GvHD (Przepiorka D, et al)

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a hematological malignancy or aplastic anemia (AA) and is undergoing a first allogeneic transplant procedure.
2. Meet one of the following underlying disease criteria:

   a. Acute myelogenous leukemia (AML) i. First or subsequent morphologic remission b. Acute lymphoblastic leukemia (ALL) i. First or subsequent morphologic remission c. Chronic myelogenous leukemia (CML) i. Chronic phase; or ii. Accelerated phase d. Multiple Myeloma (MM) i. Not more than 20% plasma cells in the bone marrow e. Myelodysplastic syndrome (MDS), including chronic myelomonocytic leukemia (CMML), who have received at least one previous induction regimen and have <10% blasts f. Myeloproliferative disorder (MPD), including; i. myeloid metaplasia, and ii. myelofibrosis g. Non-Hodgkin's Lymphoma (NHL) i. High-risk NHL in first remission; or ii. Relapsed or refractory NHL h. Hodgkin's lymphoma (HL) beyond first remission i. Aplastic anemia (AA)
3. Male or female, age ≥18 years of age
4. Reasonable expectation of survival for at least 3 months, if the transplant procedure is successful
5. Eastern Cooperative Oncology Group (ECOG) status of 0-2 or Karnofsky Performance Status (KPS) of > 60
6. Transplant Donor

   1. Part 1 (Phase 1: Dose Escalation Phase):

      Unrelated transplant donor with no more than 1 HLA allele or antigen mismatch, defined as loci A, B, C and DR (note: DQ is excluded)
   2. Part 2 (Phase 2a: Expansion Phase):Related or unrelated transplant donor, with no more than 1 HLA allele or antigen mismatch, defined as loci A, B, C and DR (note: DQ is excluded).
7. Source of the allograft

   1. Part 1 (Phase 1: Dose Escalation Phase):Unmodified (non-manipulated) bone marrow, or mobilized peripheral blood stem cell (PBSC) transplant, using G-CSF as the mobilizing agent.
   2. Part 2: (Phase 2a: Expansion Phase) Unmodified (non-manipulated) bone marrow, or mobilized peripheral blood stem cell (PBSC) transplant, using G-CSF as the mobilizing agent.
8. Anti-graft-versus-host disease (GvHD) prophylaxis:

   A calcineurin inhibitor [either tacrolimus (FK506) or cyclosporin A)], in combination with either methotrexate (MTX), mycophenolate mofetil (MMF) or sirolimus (RAPA) all at doses as per the institutional protocols
9. Adequate hepatic function, with bilirubin not exceeding the upper limit of normal (except when attributed to Gilbert's Disease), and AST and ALT of less than 1.5 times the upper limit of normal
10. No clinically significant cardiac conduction disorder on screening ECG
11. Serum creatinine ≤ 2.0 mg/dL
12. Female patients of childbearing potential must have a negative serum pregnancy test prior to enrollment and must agree to use dual method of contraception for 30 days after study drug administration. Approved methods of contraception include, an IUD with spermicide, a female condom with spermicide, a diaphragm with spermicide, a cervical cap with spermicide, use of a condom with spermicide by sexual partner or a sterile sexual partner.
13. If male, subjects must be sterile or willing to use an approved method of contraception from the time of Informed Consent to 30 days after study drug treatment. Males must be willing to refrain from sperm donation within 30 days after study drug treatment.
14. No clinically significant acute or chronic medical condition that in the opinion of the investigator will interfere with study participation
15. No clinically significant laboratory abnormalities as determined by the Principal Investigator, in consultation with the Sponsor's Medical Monitor
16. No active infection
17. Have signed written informed consent before undergoing any study related procedures and is willing to comply with all study procedures

Exclusion Criteria:

1. Female subjects who are pregnant or lactating
2. Subjects about to undergo a non-ablative or non-myeloablative transplant
3. AML or ALL patient who are in relapse (>5% blasts) or who are defined as primary refractory
4. Blast crisis CML
5. Radiation, chemotherapy, immunotherapy in the previous 3 weeks, unrelated to the transplant procedure
6. Subjects who, in the judgment of the Investigator have not recovered from the effects of previous therapy
7. Subject who is about to undergo cord blood transplantation
8. Procedures that are intended to deplete regulatory T-cells from donor transplant materials
9. Known or suspected HIV infection
10. Active hepatitis A, B, or C infection in recipient or donor
11. Uncontrolled active infection requiring IV antibiotics in recipient or donor
12. Major surgery within 1 month before Day 0
13. Participation in an investigational study within 1 month prior to Day 0
14. Prior treatment with anti-CD3 antibodies
15. Treatment with anti-CD20 antibodies or anti-thymocyte globulin (ATG) within 3 months of the AHSCT procedure (i.e. infusion of transplant material and RGI-2001).
16. Vaccination within the preceding 2 weeks prior to the planned dose of RGI-2001
17. Planned vaccination within 2 months after study drug administration
18. Known history of cardiac dysfunction (e.g. <50% ejection fraction), ischemia, conduction abnormalities, or myocardial infarction in the previous six months
19. Cardiac pacemaker or automatic implantable cardioverter-defibrillator
20. Marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms
21. Congenital long QT syndrome or family history of long QT syndrome
22. History of additional risk factors for torsades de pointes (TdP) (e.g., heart failure, hypokalemia)
23. Bundle branch block
24. Connective tissue/rheumatologic disorders
25. History of autoimmune disease
26. History of solid tumor, excluding non-melanoma skin or cervical carcinoma after curative resection, within the preceding 5 years
27. Uncontrolled diabetes
28. Prior allogeneic hematopoietic stem cell transplantation
29. Any other prior organ transplant
30. Psychiatric or addictive disorders that preclude obtaining reliable informed consent
31. Any other condition that, in the opinion of the investigator, renders the subject unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) or maximum feasible dose (MFD) of RGI-2001 | By day 29
  The primary outcome measures are:
  * The incidence and severity of adverse events
  * The maximum tolerated dose (MTD) or maximum feasible dose (MFD) of RGI-2001, administered as a single intravenous infusion approximately 30 minutes after AHSCT

SECONDARY OUTCOMES:
Pharmacodynamic Effects | Within 100 days from AHSCT
  Evaluate biomarkers to assess the potential pharmacodynamic effects of RGI-2001 through biomarkers and cytokine assessments. Exploratory biomarkers for efficacy in reducing GvHD include IL-2R, TNFR1, HGF. Cytokines will be evaluated for both safety and for evidence of mechanism of action and include IL-2, IL-4, IL-6, IL-8, IL-10, IL-12, MIG, TNF-α and IFN-γ.
Pharmacokinetics of RGI-2001 | Within first 8 days
  Obtain pharmacokinetic parameters such as Cmax, Cmin, Tmax, AUC and half-life of the study drug in plasma.
Efficacy in reducing the intensity of GvHD | Within the first 100 days after AHSCT
  The time to onset, peak intensity and course of GvHD after the AHSCT procedure will be monitored according to the Modified Keystone Criteria for Acute Graft-Versus-Host Disease.
Optimal Dose of RGI-2001 | Within first 100 days after AHSCT
  Determine optimal doses of RGI-2001 for further evaluation based on pharmacodynamic response and effectiveness in reducing the intensity of GvHD

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCSD Moores Cancer Research Institute, San Diego, California
  - Stanford School of Medicine, Stanford, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Ohio State University Comprehensive Cancer Center - The James, Columbus, Ohio
  - Methodist Healthcare System, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- See also: Regimmune Company Website — http://www.regimmune.com
- See also: Fred Hutchinson Cancer Research Center — http://www.fhcrc.org
- See also: Stanford School of Medicine — http://med.stanford.edu
- See also: UCSD Moores Cancer Center — http://cancer.ucsd.edu/Pages/default.aspx
- See also: OSU The James Comprehensive Cancer Center — http://cancer.osu.edu/Pages/index.aspx